CLINICAL TRIAL: NCT04856046
Title: Detection of Plasma DNA Methylation in Peripheral Blood From Patients With Hepatocellular Carcinoma (ATHENA)
Brief Title: Detection of Plasma DNA Methylation in Peripheral Blood From Patients With Resectable Liver Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-000878; NCI-2021-02991 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-14; First posted 2021-04-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Resectable Hepatocellular Carcinoma
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical record review): Patients undergo collection of blood samples at 4-6 weeks prior to surgery/ablation and at 12 weeks, 6, 12, 18 and 24 months after surgery/ablation. Patients' previously collected tissue samples are analyzed. Patients' medical records are also reviewed at baseline, 4-6 weeks prior to surgery/ablation, 12 weeks, 6, 12, 18 and 24 months after surgery/ablation, and then every 6 months for 3 years.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study explores the potential values of a new blood test approach to detect measurable residual disease or early coming back of cancer (recurrence)/cancer growing, spreading, or getting worse (progression) in patients with liver cancer that can be removed by surgery (resectable). The development of novel cancer biomarkers for liver cancer may help in clinical decision making and lead to improvements in patient outcomes by facilitating prediction of the response to specific treatments, improved monitoring of patients on treatment, and better prognostication of patient outcomes, thus improving stratification for clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To isolate plasma deoxyribonucleic acid (DNA) methylation panel from the peripheral blood of treated patients with hepatocellular carcinoma that will correlate with disease progression or measurable residual disease.

II. To correlate the mutations/ DNA methylation in peripheral blood with those identified in parallel tumor samples from the same patients with hepatocellular (HCC).

OUTLINE:

Patients undergo collection of blood samples at 4-6 weeks prior to surgery/ablation and at 12 weeks, 6, 12, 18 and 24 months after surgery/ablation. Patients' previously collected tissue samples are analyzed. Patients' medical records are also reviewed at baseline, 4-6 weeks prior to surgery/ablation, 12 weeks, 6, 12, 18 and 24 months after surgery/ablation, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has planned resection or ablation of suspected hepatocellular carcinoma
* Patient is classified as resectable T1/T2 hepatocellular carcinoma (HCC) (solitary tumors less than or equal to 2 cm OR solitary tumors without vascular invasion > 2cm or solitary tumor with vascular invasion > 2cm, or multiple tumors, none > 5cm) OR BCLC stage A (Single lesion of ANY size or 3 nodules or less with each being 3cm or less)

Exclusion Criteria:

* Patient is younger than 18 years of age
* Females who are pregnant or attempt to become pregnant
* Patient with significant anemia (hemoglobin [Hb] < 7g/dL)
* Patient has known cancer outside of the liver 5 years prior to current blood collection (not including basal cell or squamous cell skin cancers)
* Patient has had a biopsy to the target organ and/or lesion within 3 days before blood collection
* Patient has had an intervention to completely remove current target pathology
* Target pathology is a recurrence of previously treated HCC
* Patient has had prior resection or ablation for target lesion
* Patient has had prior or active chemotherapy or radiation for target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Multi-target hepatocellular carcinoma panel (MHP) score | Up to 1 year
  Descriptive statistics will be used. The association between the MHP score and patient and tumor characteristics with state occupancy probability will be examined using the Cox proportional hazards model. Serial measurements of the MHP score obtained on subsequent visits will be accounted for within the Cox model by treating them as time varying covariate. To assess the relative importance of the MHP score to individual alpha fetoprotein (AFP) levels for the prediction of hepatocellular carcinoma recurrence, the area under the receiver operator characteristic curve will be compared between the MHP score model and an AFP only model.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen H. Tran, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials